CLINICAL TRIAL: NCT00478946
Title: A Phase I Open-Label Study of Picoplatin in Combination With 5-Fluorouracil and Leucovorin as Initial Therapy in Subjects With Metastatic Colorectal Cancer
Brief Title: A Study of Picoplatin in Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Poniard Pharmaceuticals (Industry)
Responsible Party: Robert Earhart, MD, PhD, Poniard Pharmaceuticals
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0501
Record Dates: First submitted 2007-05-23; First posted 2007-05-25 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; picoplatin; FOLFOX; FOLPI; chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — amminedichloro(2-methylpyridine)platinum(II); Fluorouracil; Leucovorin; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Picoplatin, 150 mg/m2, 5-FU and leucovorin (q 4 weeks, Schedule B). Leucovorin, 400 mg/m2 in D5W and leucovorin (± picoplatin) will be followed by a 5-FU bolus of 400 mg/m2 and then by 5-FU, 2,400 mg/m2 in D5W administered as a 46-hour continuous infusion.
  Interventions: Drug: (FOLPI) Picoplatin with 5-FU and Leucovorin; Drug: FOLPI
- 2 (Active Comparator): FOLFOX Oxaliplatin 85 mg/m2, as a 2-hour infusion Leucovorin (400 mg/m2 in D5W) and Oxaliplatin. Leucovorin + oxaliplatin will be followed by a 5-FU bolus of 400 mg/m2 and then by 5-FU, 2400 mg/m2 in D5W administered as a 46-hour continuous infusion.
  Interventions: Drug: FOLFOX

INTERVENTIONS:
Drug: (FOLPI) Picoplatin with 5-FU and Leucovorin — Picoplatin, 150 mg/m2, 5-FU and leucovorin (q 4 weeks, Schedule B). Leucovorin, 400 mg/m2 in D5W and leucovorin (± picoplatin) will be followed by a 5-FU bolus of 400 mg/m2 and then by 5-FU, 2,400 mg/m2 in D5W administered as a 46-hour continuous infusion.
  Arms: 1
Drug: FOLPI — Picoplatin, 150 mg/m2 to be administered with every alternate cycle of 5-FU and leucovorin (q 4 weeks, Schedule B). Leucovorin, 400 mg/m2 in D5W, will be administered as a 2-hour infusion, either alone or, if the patient is to receive picoplatin that cycle, at the same time as picoplatin, in separate bags using a Y-line. The leucovorin (± picoplatin) will be followed by a 5-FU bolus of 400 mg/m2 and then by 5-FU, 2,400 mg/m2 in D5W administered as a 46-hour continuous infusion.
  Arms: 1
Drug: FOLFOX — Oxaliplatin 85 mg/m. Leucovorin (400 mg/m2 in D5W). Oxaliplatin and leucovorin Leucovorin + oxaliplatin 5-FU bolus of 400 mg/m2 and then by 5-FU, 2400 mg/m2 in D5W administered as a 46-hour continuous infusion.
  Arms: 2

SUMMARY:
Colorectal cancer is a type of cancer that begins in the large intestine (colon) or the rectum (end of the colon). Several drugs are often given in combination to treat colorectal cancer. One of the most active treatment combinations is known as FOLFOX, which is a combination of 5-fluorouracil (5-FU), leucovorin, and oxaliplatin. Oxaliplatin is a type of platinum drug and was approved by the FDA in 2004. While generally well-tolerated, oxaliplatin may cause toxicity to the nerves, such as sensory loss or cold sensitivity.

Picoplatin is a new type of platinum drug that has shown activity with 5-FU in pre-clinical studies and has undergone extensive Phase 1 and Phase 2 testing in a variety of cancers. No significant nerve toxicity has been seen in previous studies of picoplatin.

This study will review the safety and effectiveness of FOLPI, which is the combination of 5-FU and leucovorin with picoplatin in participants with colorectal cancer.

DETAILED DESCRIPTION:
Subjects will be randomized centrally to treatment with picoplatin administered either every two or every four weeks and will be assigned a dose of picoplatin dependent on the study results to date. Each patient will also receive therapy every two weeks with 5-FU and leucovorin. In each schedule, the cohort size will be 3 subjects, to be expanded to 6 subjects if a dose-limiting toxicity is observed. If not dose-limiting toxicity observed among the 3 subjects within a cohort, picoplatin dose escalation may proceed, until the maximum tolerated dose is established.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the colon or rectum.
* Metastatic disease consistent with colorectal adenocarcinoma. Stage M1, and not amenable to curative surgery. Subjects with only locally persistent or only locally recurrent disease are not eligible.
* No prior systemic therapy for metastatic cancer. Prior adjuvant chemotherapy with a 5-FU-based treatment regimen not containing oxaliplatin or irinotecan is acceptable after a treatment-free interval of at least 6 months.
* ECOG performance score (PS) of 0 or 1.
* Life expectancy more than 3 months.
* Subject must have measurable disease, defined by the RECIST criteria.
* At least 28 days must have elapsed since prior surgery except venous access device placement.
* At least 28 days must have elapsed since prior radiotherapy.
* At least 28 days must have elapsed since a prior investigational agent.
* Absolute neutrophil count (ANC) equal to or greater than 1.5 x 10^9/L.
* Platelet count equal to or greater than 100 x 10^9/L.
* Hemoglobin equal or greater than 10g/dL (must be obtained at least 3 days after any transfusion).
* Serum AST and ALT levels less than or equal to 2.5 times upper limit of normal (ULN) or less than 5 times ULN if liver involvement is present.
* Serum bilirubin of less than or equal to 1.5 ULN.
* Serum creatinine of less than or equal to ULN.
* Women of childbearing potential must have a negative pregnancy test (serum or urine beta HCG).
* All subjects must agree to use appropriate birth control methods while on study and for 1 month after completion of study chemotherapy.

Exclusion Criteria:

* Concurrent use of EGFR inhibitors or anti-VEGF agents.
* No clinically significant obstructive symptoms or intestinal bleeding.
* Significant chronic or recent acute gastrointestinal disorder with diarrhea as a major symptom (e.g. Crohn's disease, ulcerative colitis, malabsorption syndrome, Grade 2+ diarrhea of any etiology at baseline).
* History of serious cardiac disease, defined as myocardial infarction within six months of enrollment, congestive heart failure classified by the New York Heart Association as class III or IV, uncontrolled cardiac arrhythmias, poorly controlled or unstable angina, or electrocardiographic evidence of acute ischemia.
* Clinical evidence of brain metastases or central nervous system disease.
* Symptomatic peripheral neuropathy (equivalent to Grade 2 or higher CTCAE toxicity criteria).
* Uncontrolled intercurrent illness (e.g. active infection).
* Pregnant or nursing.
* Serious medical or psychiatric illness that could potentially interfere with the completion of study treatment according to this protocol.
* Malignancy other than colorectal carcinoma within the past 5 years, except, curatively treated, superficial skin cancer or carcinoma in situ of the cervix or breast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2006-04; Primary Completion 2009-12 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
dose-limiting toxicity | within the first four weeks of treatment
maximum tolerated dose | within the first two cycles of treatment

SECONDARY OUTCOMES:
safety and efficacy | duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Robert Earhart, MD, PhD, Study Director — Poniard Pharmaceuticals
Locations (16):
- Russia (16):
  - Leningrad Regional Oncology Center, Chemotherapy Department - Phase 2, Kuzmolovsky Village, Vsevolozhsk
  - Regional Oncology Center - Phase 2, Astrakhan
  - Chelyabinsk Regional Oncology Center - Phase 1, Chelyabinsk
  - Regional Oncology Center, Chemotherapy Department - Phase 2, Engel's
  - Kazan Oncology Center, Kazan'
  - Blokhin Russian Oncology Research Center - Phase 1, Moscow
  - Semashko Central Clinical Hospital #2 - Phase 1, Moscow
  - Medical Radiology Research Center of Russian Academy of Medical Sciences- Phase 1, Obninsk
  - Republic Oncology Center of the Ministry of Healthcare of Karelia Republic - Phase 2, Petrozavodsk
  - Rostov Research Institute of Oncology- Phase 2, Rostov-na-Dony
  - St. Petersburg Academy of Postgraduate Education - Phase 2, Saint Petersburg
  - St. Petersburg Mechnikov State Medical Academy - Phase 2, Saint Petersburg
  - St. Petersburg City Oncology Center - Phase 1, Saint Petersburg
  - Regional Clinical Oncology Center - Phase 2, Ulyanovsk
  - Voronezh Regional Clinical Oncology Center - Phase 2, Voronezh
  - Yaroslavl Regional Oncology Center - Phase 1, Yaroslavl

REFERENCES:
- [Background] Douillard JY, Schiller J. ZD0473 combined with other chemotherapeutic agents for the treatment of solid malignancies. Eur J Cancer. 2002 Dec;38 Suppl 8:S25-31. doi: 10.1016/s0959-8049(02)80020-x. PMID 12645909
- [Background] Beale P, Judson I, O'Donnell A, Trigo J, Rees C, Raynaud F, Turner A, Simmons L, Etterley L. A Phase I clinical and pharmacological study of cis-diamminedichloro(2-methylpyridine) platinum II (AMD473). Br J Cancer. 2003 Apr 7;88(7):1128-34. doi: 10.1038/sj.bjc.6600854. PMID 12671715
- [Background] Raynaud FI, Boxall FE, Goddard PM, Valenti M, Jones M, Murrer BA, Abrams M, Kelland LR. cis-Amminedichloro(2-methylpyridine) platinum(II) (AMD473), a novel sterically hindered platinum complex: in vivo activity, toxicology, and pharmacokinetics in mice. Clin Cancer Res. 1997 Nov;3(11):2063-74. PMID 9815598
- [Background] Holford J, Raynaud F, Murrer BA, Grimaldi K, Hartley JA, Abrams M, Kelland LR. Chemical, biochemical and pharmacological activity of the novel sterically hindered platinum co-ordination complex, cis-[amminedichloro(2-methylpyridine)] platinum(II) (AMD473). Anticancer Drug Des. 1998 Jan;13(1):1-18. PMID 9474239
- [Background] Holford J, Sharp SY, Murrer BA, Abrams M, Kelland LR. In vitro circumvention of cisplatin resistance by the novel sterically hindered platinum complex AMD473. Br J Cancer. 1998;77(3):366-73. doi: 10.1038/bjc.1998.59. PMID 9472630
- [Background] Rogers P, Boxall FE, Allott CP, Stephens TC, Kelland LR. Sequence-dependent synergism between the new generation platinum agent ZD0473 and paclitaxel in cisplatin-sensitive and -resistant human ovarian carcinoma cell lines. Eur J Cancer. 2002 Aug;38(12):1653-60. doi: 10.1016/s0959-8049(02)00107-7. PMID 12142057
- [Background] Sharp SY, O'Neill CF, Rogers P, Boxall FE, Kelland LR. Retention of activity by the new generation platinum agent AMD0473 in four human tumour cell lines possessing acquired resistance to oxaliplatin. Eur J Cancer. 2002 Nov;38(17):2309-15. doi: 10.1016/s0959-8049(02)00244-7. PMID 12441268
- [Background] Plasencia C, Abad A, Martinez-Balibrea E, Taron M. Antiproliferative effects of ZD0473 (AMD473) in combination with 5-fluorouracil or SN38 in human colorectal cancer cell lines. Invest New Drugs. 2004 Nov;22(4):399-409. doi: 10.1023/B:DRUG.0000036682.99818.71. PMID 15292710
- [Background] Murakami H, Tamura T, Yamada Y, Yamamoto N, Ueda Y, Shimoyama T, Saijo N. ZD0473 pharmacokinetics in Japanese patients: a Phase I dose-escalation study. Eur J Cancer. 2002 Dec;38 Suppl 8:S1-5. doi: 10.1016/s0959-8049(02)80012-0. PMID 12645906